CLINICAL TRIAL: NCT01591889
Title: A Single Dose, Two-Period, Two-Treatment, Two-Way Crossover Bioequivalence Study of Tinidazole 500 mg Tablets Under Fed Conditions
Brief Title: Crossover Bioequivalence Study of Tinidazole 500 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Sponsor
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TINI-T500-PVFD-1
Record Dates: First submitted 2012-05-01; First posted 2012-05-04 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Trichomoniasis
MeSH Terms: conditions — Trichomonas Infections | interventions — Tinidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- tindamax (Active Comparator): 500 mg tablet
  Interventions: Drug: Tinidazole
- tinidazole (Active Comparator): 500 mg tablet
  Interventions: Drug: Tinidazole

INTERVENTIONS:
Drug: Tinidazole — 500 mg tablet
  Other Names: Tindamax®
  Arms: tindamax
Drug: Tinidazole — 500 mg tablet
  Other Names: Tindamax
  Arms: tinidazole

SUMMARY:
The objective of this study was to prove the bioequivalence of Roxane Laboratories' Tinidazole 500 mg Tablet under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to tinidazole or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, MD, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States